CLINICAL TRIAL: NCT05001061
Title: Sublingual vs Vaginal Misoprostol for Termination of First Trimesteric Missed Abortion
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mahmoud Emam Ahmed, Resident in obstetrics and gynecology, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Misoprostol abortion
Record Dates: First submitted 2021-08-02; First posted 2021-08-11 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Missed Abortion
MeSH Terms: conditions — Abortion, Missed | interventions — Misoprostol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sublingual Misoprostol for termination of first trimester missed abortion (Active Comparator): Patients diagnosed as first trimester missed abortion will receive sublingual Misoprostol 800 micrograms every 4 hours up to five doses
  Interventions: Drug: Misoprostol Pill
- Vaginal Misoprostol for termination of first trimester missed abortion (Active Comparator): Patients diagnosed as first trimester missed abortion will receive vaginal Misoprostol 800 micrograms every 4 hours up to five doses
  Interventions: Drug: Misoprostol Pill

INTERVENTIONS:
Drug: Misoprostol Pill — sublingual versus vaginal Misoprostol in termination of first trimester missed abortion

SUMMARY:
Efficacy of sublingual versus vaginal misoprostol in termination of first trimester missed abortion

DETAILED DESCRIPTION:
study will be made on female patients with first trimester missed abortion confirmed by ultrasound . Participants will be divided into 2 groups one group (A) will receive sublingual Misoprostol and the other group(B) will receive vaginal Misoprostol as a 800 micro grams every 4 hours in both groups up to five doses the aim of the study is to compare efficay of sublingual and vaginal Misoprostol in complete termination of first trimester missed abortion and which route is the best will less side effects.

ELIGIBILITY:
Inclusion Criteria:

* Women with an ultrasound diagnosis of missed abortion < 13 weeks gestation without any clinical criteria of Inevitable abortion.

Exclusion Criteria:

* Patients refused the medical treatment.
* Patients have contraindications of the drug (Misoprostol).
* Missed abortion associated with any signs of sepsis

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 288 (Estimated)
Dates: Start 2021-08-03 (Estimated); Primary Completion 2021-10-15 (Estimated); Study Completion 2021-10-16 (Estimated)

PRIMARY OUTCOMES:
The occurance of complete abortion within 24 hours with Misoprostol drug | Within 24 hours
  Efficacy of sublingual and vaginal Misoprostol in complete termination of first trimester missed abortion
Which route is the best and less side effects in complete termination of first trimester missed abortion by Misoprostol drug | within 24 hours
  Vaginal versus sublingual route of administration of Misoprostol for complete termination of first trimester missed abortion

REFERENCES:
- [Background] Allameh Z, Goharian M, Eslamian M. Effect of misoprostol with and without letrozole on the induction of abortion for women with first-trimester missed abortion. Int J Gynaecol Obstet. 2020 Nov;151(2):214-218. doi: 10.1002/ijgo.13326. Epub 2020 Sep 1. PMID 32700359
- [Background] Tang OS, Gemzell-Danielsson K, Ho PC. Misoprostol: pharmacokinetic profiles, effects on the uterus and side-effects. Int J Gynaecol Obstet. 2007 Dec;99 Suppl 2:S160-7. doi: 10.1016/j.ijgo.2007.09.004. Epub 2007 Oct 26. PMID 17963768